CLINICAL TRIAL: NCT06698666
Title: The Efficacy of Statins in Management of Major Depression Disorder (MDD) Among Adult Patients Attending the Outpatient Clinics of El Demerdash Hospital.
Brief Title: Efficacy of Statins Among Major Depressive Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Silvana Nader, Assisstant lecturer, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 187/2022
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder; MDD
Keywords: Rosuvastatin; Major depressive disorder; MADRS scale
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Rosuvastatin Calcium; Tablets; Sertraline

STUDY DESIGN:
Intervention Model Description: - Study Interventions The study is a 12-week, parallel group, randomised controlled trial (RCT) in participants with mild to moderate MDD. A baseline line assessment will be done by obtaining the socio-demographic data for the whole participants and The participants will be allocated into either groups First Group:Participants will receive Selective Serotonin Reutake Inhibitors (SSRI)(Sertraline).
  Second Group:Participants will receive Selective Serotonin Reutake Inhibitors (SSRI) (Sertraline) and rosuvastatin 10 mg/day.
  Assessments will be scheduled at baseline and weeks 4, 8, and 12. Randomisation and Blinding: Participants will be allocated into either 2 groups: control group (SSRI only) or interventional group (SSRI plus statins) randomly by giving them sealed envelopes containing code for control or interventional group Interventions: The participant will be randomly assigned to the interventional, or control group on a 1:1 basis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Control Group (Other): The Control Group will receive the standard treatment of depression including SSRI (Sertraline) only
- The Interventional group (Experimental): the interventional group will receive the standard treatment of depression including SSRI (Sertraline) in addition to the10 mg/day rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin 10 mg tablet. — The dose of rosuvastatin was derived from literature describing the doses at which the agents' targeted actions are effective and safe. The 10- mg rosuvastatin dose reflects the lowest prescribed therapeutic dose A serum cholesterol level will be drawn from the whole participants and sent to the central laboratories of El-Demerdash hospital at baseline and at week 12.
  At each visit, participants will be requested to return all unused investigational products. Adherence to medication will be assessed by a pill count.
Drug: Sertraline Pill — Both control and intervention group will receive the sertraline as a standard therapy

SUMMARY:
The goal of this clinical trial is to learn if drug Rosuvastatin 10 mg works to treat MDD in adults. It will also learn about the safety of Rosuvastatin 10 mg .The main questions it aims to answer are:

Does Rusovastatin lower the score of The Montgomery Asberg Depression Rating Scale (MADRS) among adult participants with Major Depression Disorder ( MDD )? What medical problems do participants have when taking drug ABC?

Participants will:

Take Rosuvastatin 10 mg every day for 3 months Visit the clinic once every 4 weeks for checkups and tests Report any side effects for Rosuvastatin 10 mg and reassess the severity of depression using The Montgomery Asberg Depression Rating Scale (MADRS)

DETAILED DESCRIPTION:
* Type of Study: Randomised Controlled Trial (RCT)
* Study Setting: Psychiatry institute of Professor Ahmed Okasha, El- Demerdash hospitals.
* Study Period: starting from September 2022 till completion of sample size
* Study Population

Any adult patient aged 20 -45 years old attending the psychiatric clinic at the Psychiatry institute of Professor Ahmed Okasha, El- Demerdash hospitals with mild or moderate depression.

Diagnostic criteria for minor depression according to the American Psychiatric Association's Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)

We diagnose minor depressive episodes according to all of the following criteria (A through F).

A. Two to four of the following symptoms have been present during the same two-week period:

1. Dysphoria - Depressed mood most of the day, nearly every day
2. Anhedonia - Markedly diminished interest or pleasure most of the day, nearly every day
3. Significant appetite or weight change
4. Insomnia or hypersomnia nearly every day
5. Psychomotor agitation or retardation (observable by others)
6. Anergia - Fatigue nearly every day
7. Thoughts of worthlessness or inappropriate guilt nearly every day
8. Impaired concentration or memory nearly every day
9. Recurrent thoughts of death or suicide, or suicide attempt

B. At least one of the symptoms includes dysphoria or anhedonia C. The symptoms cause clinically significant distress of psychosocial impairment D. The symptoms are not due to the physiologic effects of a substance, medication, or general medical condition E. Persistent depressive disorder (dysthymia) and cyclothymic disorder are not present F. The mood disturbance does not occur exclusively during a psychotic disorder

* Sampling Method: Convenience sample
* Sample Size

Using G power software for sample size calculation, setting power at 80% and alpha error at 0.05, it is estimated that sample size of 65 patients per group will be needed to detect a statistical difference between two groups regarding MADRS score after 12 weeks assuming medium effect size, difference between two groups (Cohen's coefficient = 0.5.

Assuming 10% dropout rate, sample size of 72 participants per group will be needed.

Ethical Considerations

1. Approval from the research ethical committee of Faulty of Medicine Ain Shams University will be taken.
2. An informed consent will be used to inform the participants about all the steps of the study and the risks and benefits of the study.
3. Anonymous questionnaires will be used to assure confidentiality of the data. Regarding the Confidentiality of data, the Principle investigator and Co -investigator will be the only persons having access to the patient's data.

Study Tools

* First, a baseline line assessment will be done by obtaining the socio-demographic data (including age, gender, level of education, occupation, marital status, residence and family history of any psychiatric illness ) for the whole participants
* Second, diagnosis of major depressive disorder will be confirmed using the Structured Clinical Interview for DSM-IV Axis I Disorders, patient version (SCID-I/P)

The Structured Clinical Interview for DSM-4-Clinician Edition is a screening procedure used to diagnose DSM-4 Axis I disorders (major psychiatric disorders). It comprises seven diagnostic modules based on various diagnostic groups: mood disorders, depression, drug abuse, anxiety, somatoform disorders, eating disorders, and adjustment disorders. El-Missiry translated the SCID-I-CV into Arabic in 2004, and its use was confirmed in various studies performed in Egyptian study centers.

- Third, severity of depression will be determined using the Montgomery Asberg Depression Rating Scale (MADRS) including those who are between 7 and 34.

* The Montgomery Asberg Depression Rating Scale (MADRS) is used by clinicians to assess the severity of depression among patients with a diagnosis of depression. It is designed to be sensitive to change resulting from antidepressant therapy.
* Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
* The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts

Usual cutoff points are:

* 0 to 6 - normal /symptom absent
* 7 to 19 - mild depression
* 20 to 34 - moderate depression
* >34 - severe depression.

  · Time: Interviews take 20 to 60 minutes to complete.

  · Subscales: The MADRS has 10 subtests (each item is therefore considered a subtest): 1. Apparent sadness; 2. Reported sadness; 3. Inner tension; 4. Reduced sleep; 5. Reduced appetite; 6. Concentration difficulties; 7. Lassitude; 8. Inability to feel; 9. Pessimistic thoughts; 10. Suicidal thoughts

  · Equipment: Only the questionnaire and a pencil are required to complete the MADRS.

  · Training: No formal training is required to complete the MADRS.
* Fourth, serum cholesterol level will be drawn and sent to the central laboratories of El-Demerdash hospital at baseline and at week 12.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 45 years;
* diagnosis of current MDD, verified using the Structured Clinical Interview for DSM-IV Axis I Disorders, patient version (SCID-I/P);
* The Montgomery Asberg Depression Rating Scale (MADRS) score of 7 to 34, indicating mild to moderate depression;
* the ability to give informed consent and to comply with standard procedures;
* Males and females; and
* Stable pharmacological treatment for at least 2 weeks prior to enrolment (changes to medication dose or frequency of therapy excepted) if currently being treated.

Exclusion Criteria:

* lifetime or current SCID-I/P diagnosis of a psychotic disorder;
* lifetime SCID-I/P diagnosis of bipolar I or II disorder or alcohol dependence;
* acute or unstable systemic medical disorder;
* inability to comply with the requirements of informed consent or the study protocol;
* history of intolerance or allergy to study medications;
* Current pregnancy or breast feeding;
* Current regular use of statins, corticosteroids, or any other immunomodulatory agents; and
* Females on Contraception.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of depression among Participants with MDD as Assessed by MADRS scale | 3 months (12 weeks)
  Severity of depression will be determined using the Montgomery Asberg Depression Rating Scale (MADRS) including those who are between 7 and 34.
  * The Montgomery Asberg Depression Rating Scale (MADRS) is used by clinicians to assess the severity of depression among patients with a diagnosis of depression. It is designed to be sensitive to change resulting from antidepressant therapy.
  * Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  * The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts
  * Time:
  Interviews take 20 to 60 minutes to complete.

CONTACTS AND LOCATIONS:
Locations (1):
- El demerdash hospital, Cairo, Al Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No